CLINICAL TRIAL: NCT04467229
Title: Early Detection of Mental Disorders in Adolescents With Chronic Pain: Creation of a Screening Tool for Use by the General Practitioner
Acronym: REPERADO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200623
Record Dates: First submitted 2020-05-25; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain; Mental Disorder
Keywords: Chronic Pain; Mental Disorders
MeSH Terms: conditions — Chronic Pain; Mental Disorders | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focus group with chronically painful adolescents (Experimental): Adolescents with chronic pain
  Interventions: Behavioral: Focus group

INTERVENTIONS:
Behavioral: Focus group — 5 to 10 adolescents will participate in a discussion group lead by a paediatrician and a psychologist from the Centre de la Douleur de Trousseau. Two groups will be organized, the length of the group discussion being one hour. These focus groups will explore the adolescents' perception of the questionnaire and of different elements of the screening. The group will undergo full transcription. The verbatim will be anonymous and will be analysed through qualitative methods.

SUMMARY:
This research aims to create a tool for detection of mental health disorders in adolescents with chronic pain. The first part is testing a screening questionnaire and comparing in with existing questionnaires. The second part involves two focus group with the adolescents aimed at recording their perception of the questionnaire.

DETAILED DESCRIPTION:
First part : creation of a screening tool. After detailed interviews with chronic pain experts and bibliographic research, a screening tool for mental disorders in chronically painful adolescents has been designed for use by the general practitioner. This tool is composed of 10 questions, making up a score of 10 points. The tool will be compared to two screening tools used in different clinical contexts, the HAD scale and the RPPS scale, in order to determine a positivity threshold. There is only one center participating in the research, the Centre de la Douleur et de la migraine de l'hôpital Trousseau (Trousseau Hospital Pain Center). Parents' consent is required for participation. For this assessment, the adolescents (between 10 and 18 years old) that see a doctor at the Centre de la douleur, will be asked to fill up the questionnaires in the waiting room. The filling of the questionnaire takes a few minutes. At the end of the appointment, the doctor will read the questionnaire to check that all elements have been addressed during the appointment.

Second part : focus group on the questionnaire: 5 to 10 adolescents will participate in a discussion group lead by a paediatrician and a psychologist from the Centre de la Douleur de Trousseau. Two groups will be organized, the length of the group discussion being one hour. These focus groups will explore the adolescents' perception of the questionnaire and of different elements of the screening. The group will undergo full transcription. The verbatim will be anonymous and will be analysed through qualitative methods.

The data will help designing a guidebook for the clinician explaining the main points in screening for mental disorders in chronic pain adolescent patients.

A validation study for the screening tool will be eventually carried out after the completion of this preliminary study.

ELIGIBILITY:
Inclusion Criteria:

* patient from 10 to 18 years old
* chronic pain (existing for more than 3 months or longer than tissue repair time)
* first consultation in the service
* Collection of the written consent of the holders of parental authority and agreement of the adolescent
* Adolescents able to understand the questionnaire and the purpose of the study
* Affiliation to a social security scheme or beneficiary

Exclusion Criteria:

Exclusion Criteria :

* Decompensated physical or psychological pathology requiring urgent medical treatment
* Heavy psychological pathology preventing the adolescent's understanding of the study
* Patient benefiting from State Medical Aid

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-06 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Screening questionnaire score | Baseline visit
  A new Screening questionnaire elaborated beforehand by the study will be answered by patients in order to detect psychological suffering in chronically painful adolescents The screening questionnaire consists in 10 items (yes/no response format)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression (HAD) score | Baseline visit
  Patients complete a Hospital Anxiety and Depression (HAD) scale questionnaire
Pediatric Pain Screening Tool (PPST) score | Baseline visit
  Patients complete a Pediatric Pain Screening Tool questionnaire
Participants feedback | up to 3 months upon recuitment
  Focus group questions will provide descriptions of patients' experiences with the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra LOISEL, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre de la douleur et de la migraine-Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No